CLINICAL TRIAL: NCT02958891
Title: Caries, Gingivitis, Dental Trauma and Fluorosis Prevalence Among IDF Recruits - an Epidemiological Survey
Brief Title: Dental Health Epidemiology Among Israel Defense Forces (IDF) Recruits
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Nirit Yavnai, Principal Investigator, Medical Corps, Israel Defense Force
Other Study IDs: 1524-2015
Record Dates: First submitted 2016-11-06; First posted 2016-11-08 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Caries, Dental; Gingivitis; Fluorosis; Dental Trauma
MeSH Terms: conditions — Dental Caries; Gingivitis; Fluoride Poisoning | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Data collection — Collection epidemiological dental measures

SUMMARY:
An epidemiological survey for prevalence description of dental morbidity (caries, gingivitis, dental trauma and fluorosis) among Israel Defense Forces (IDF) general recruits. Morbidity measures were collected from 700 recruits at their first day of military service in order to evaluate extent and burden of dental diseases among recruits. The data will enable the military dental services commanders to plan and implement dental services according to the dental needs.

DETAILED DESCRIPTION:
Caries, gingivitis, dental trauma and fluorosis epidemiological measures were collected among IDF recruits in 700 sample using short clinical evaluation without radiographs. water fluoridation ecological data will be obtained from the ministry of health. the results might impact dental services plan, professional manpower system, and the layout of the dental clinics in the IDF. It will give the professionals in the military dental services an evidence based data for planning an accurate primary and secondary prevention programs and an evaluation of dental diseases burden in order to have the "full picture" of recruits dental needs. .

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old.

Exclusion Criteria:

* Chronic bone diseases.
* Mineralization defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General IDF recruits.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
DMFT index (Decayed, Missing, Filled, Tooth) | 7 days
CPI (Community Periodontal Index) index | 7 days
TDI (Dental Trauma Index) index | 7 days
TF (Thylstrup & Fejerskov Index for dental Fluorosis) index | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Nirit Yavnai, DMD MPH, Principal Investigator — IDF Medical Corps
Locations (1):
- IDF Medical Corps, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No
Data will be published after statistical analysis only.

REFERENCES:
- [Derived] Yavnai N, Mazor S, Vered Y, Shavit I, Zini A. Caries prevalence among 18 years old, an epidemiological survey in Israel. Isr J Health Policy Res. 2020 Aug 31;9(1):45. doi: 10.1186/s13584-020-00402-4. PMID 32867853